CLINICAL TRIAL: NCT02586636
Title: Impact of OCT1 Genotype and OCT1 Inhibiting Drugs on an Individual's Tolerance of Metformin
Brief Title: Impact of OCT1 on Metformin Tolerance
Acronym: ImpOCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Dundee (Other)
Responsible Party: Principal Investigator, Laura McCreight, Principal Investigator, NHS Tayside
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2015DM13
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Tolerance
Keywords: Metformin; OCT1
MeSH Terms: interventions — Metformin; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCT1 -/- (Other): Cohort of patients with two loss of function alleles for OCT1. The participants within this group will receive metformin at increasing dose to a maximum tolerated dose over two distinct four week treatment periods. The concurrent treatment order of omeprazole and placebo will be randomised within the cohort.
  Interventions: Drug: Metformin; Drug: Omeprazole; Drug: Placebo
- OCT wt/wt (Other): Cohort of patients with two "normal" or wild type alleles for OCT1. The participants within this group will receive metformin at increasing dose to a maximum tolerated dose over two distinct four week treatment periods. The concurrent treatment order of omeprazole and placebo will be randomised within the cohort.
  Interventions: Drug: Metformin; Drug: Omeprazole; Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin is given alongside omeprazole / placebo. Started at low dose and titrated gradually over four weeks according to the individual's tolerance of metformin. We anticipate that their tolerance of metformin will be reduced by loss of function variants in OCT1, and by concurrent use of OCT1 inhibiting drugs (in our study this is omeprazole).
Drug: Omeprazole — Given as concurrent treatment in one of the two treatment periods. Omeprazole treatment dose is fixed at 20mg twice daily for four weeks duration. Omeprazole, in our study, is used as an OCT1 inhibitor, and we hypothesise that this will reduce an individual's maximum tolerated dose of metformin during concurrent treatment. This will be compared to the other treatment period in which concurrent treatment is a placebo, and therefore, the maximum tolerated dose of metformin would not be affected.
Drug: Placebo — Given as concurrent treatment in one of the two treatment periods. Placebo treatment dose is fixed at one tablet twice daily (to match the dosing pattern of omeprazole) for four weeks duration. Omeprazole, in our study, is used as an OCT1 inhibitor, and we hypothesise that this will reduce an individual's maximum tolerated dose of metformin during concurrent treatment. This will be compared to the other treatment period in which concurrent treatment is a placebo, and therefore, the maximum tolerated dose of metformin would not be affected.

SUMMARY:
Metformin is the first-line treatment for medical management of Type 2 Diabetes. Up to 25% of patients experience significant gastrointestinal symptoms and in approximate 5%, side-effects result in the discontinuation of metformin. It would be of great clinical significance if the underlying cause of this intolerance was identified.

Recent data has highlighted a metformin transporter in the gut - Organic Cation Transporter 1(OCT1) - as a potential culprit for the variability in metformin tolerance. Across a diabetic population, up to one in four people were shown to have a single reduced function allele for OCT1, with approximately 8% having two reduced function alleles. This may increase the risk of the individual experiencing metformin-associated side-effects, potentially due to accumulation within the cells lining the intestine. The investigators aim to show that loss of function of OCT1, either due to genetic variation or drug inhibition of OCT1, may lead to an increase in the symptoms associated with metformin intolerance.

The study is being undertaken at the Clinical Research Centre in Ninewells Hospital, Dundee. The investigators will recruit participants from the GoDARTS study (Genetics of Diabetes and Audit Research Tayside Study). The participants will be healthy controls, i.e. non-diabetic, and recruited according to their genotype of OCT1 (information from GoDARTS). The volunteers will then enter a matched cross-over study with two treatment periods. Metformin is taken during both treatment periods alongside either Omeprazole (a proton pump inhibitor used to prevent excess stomach acid, known to interact with OCT1) or placebo. The metformin dose is increased gradually during each period, to a maximum tolerated dose. The investigators expect to see a lower maximum tolerated dose in individuals with loss of function genotype, or in those taking concurrent omeprazole compared to placebo. The study will last approximately 9 weeks. Volunteers have 3 visits to the CRC, and weekly phone call interviews.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 80
* White European (to limit genetic variation as much as possible)
* Non-diabetic
* No previous treatment with metformin
* No known gastrointestinal pathology e.g. inflammatory bowel disease, IBS, coeliac
* No daily treatment with PPI, anti-spasmodic, or anti-motility drugs
* No daily OCT1 inhibiting drugs
* Able to complete the symptom severity score and Bristol stool chart independently i.e. no cognitive impairment or visual impairment
* Normal renal function - eGFR>60
* Known OCT1 genotype - either normal ("wild type") or two reduced function alleles.

Exclusion Criteria:

* Does not meet inclusion criteria
* Heterozygous OCT1 genotype i.e. only one reduced function allele
* Recent involvement (<30 days) in a CTIMP
* Pregnancy or planning to conceive
* Inability/unwillingness to comply with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of metformin | At the completion of the study, after approximately 1.5 years.
  Each treatment period consists of four weeks. Metformin dose titrated gradually in presence of omeprazole or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ewan R Pearson, MBBCh, PhD, Study Chair — University of Dundee / NHS Tayside
Locations (1):
- Ninewells Hospital, Dundee, Angus, United Kingdom

REFERENCES:
- [Background] Koehler MR, Wissinger B, Gorboulev V, Koepsell H, Schmid M. The two human organic cation transporter genes SLC22A1 and SLC22A2 are located on chromosome 6q26. Cytogenet Cell Genet. 1997;79(3-4):198-200. doi: 10.1159/000134720. PMID 9605850
- [Background] Koepsell H, Endou H. The SLC22 drug transporter family. Pflugers Arch. 2004 Feb;447(5):666-76. doi: 10.1007/s00424-003-1089-9. Epub 2003 Jul 19. PMID 12883891
- [Background] Han TK, Proctor WR, Costales CL, Cai H, Everett RS, Thakker DR. Four cation-selective transporters contribute to apical uptake and accumulation of metformin in Caco-2 cell monolayers. J Pharmacol Exp Ther. 2015 Mar;352(3):519-28. doi: 10.1124/jpet.114.220350. Epub 2015 Jan 6. PMID 25563903
- [Background] Proctor WR, Bourdet DL, Thakker DR. Mechanisms underlying saturable intestinal absorption of metformin. Drug Metab Dispos. 2008 Aug;36(8):1650-8. doi: 10.1124/dmd.107.020180. Epub 2008 May 5. PMID 18458049
- [Background] Muller J, Lips KS, Metzner L, Neubert RH, Koepsell H, Brandsch M. Drug specificity and intestinal membrane localization of human organic cation transporters (OCT). Biochem Pharmacol. 2005 Dec 5;70(12):1851-60. doi: 10.1016/j.bcp.2005.09.011. Epub 2005 Nov 2. PMID 16263091
- [Background] Han TK, Everett RS, Proctor WR, Ng CM, Costales CL, Brouwer KL, Thakker DR. Organic cation transporter 1 (OCT1/mOct1) is localized in the apical membrane of Caco-2 cell monolayers and enterocytes. Mol Pharmacol. 2013 Aug;84(2):182-9. doi: 10.1124/mol.112.084517. Epub 2013 May 16. PMID 23680637
- [Background] Dujic T, Zhou K, Donnelly LA, Tavendale R, Palmer CN, Pearson ER. Association of Organic Cation Transporter 1 With Intolerance to Metformin in Type 2 Diabetes: A GoDARTS Study. Diabetes. 2015 May;64(5):1786-93. doi: 10.2337/db14-1388. Epub 2014 Dec 15. PMID 25510240
- [Background] Stage TB, Brosen K, Christensen MM. A Comprehensive Review of Drug-Drug Interactions with Metformin. Clin Pharmacokinet. 2015 Aug;54(8):811-24. doi: 10.1007/s40262-015-0270-6. PMID 25943187
- [Background] Christensen MM, Brasch-Andersen C, Green H, Nielsen F, Damkier P, Beck-Nielsen H, Brosen K. The pharmacogenetics of metformin and its impact on plasma metformin steady-state levels and glycosylated hemoglobin A1c. Pharmacogenet Genomics. 2011 Dec;21(12):837-50. doi: 10.1097/FPC.0b013e32834c0010. PMID 21989078
- [Background] Christensen MMH, Hojlund K, Hother-Nielsen O, Stage TB, Damkier P, Beck-Nielsen H, Brosen K. Steady-state pharmacokinetics of metformin is independent of the OCT1 genotype in healthy volunteers. Eur J Clin Pharmacol. 2015 Jun;71(6):691-697. doi: 10.1007/s00228-015-1853-8. Epub 2015 May 5. PMID 25939711